CLINICAL TRIAL: NCT01796912
Title: Clinical Outcomes, Perfusion and Vascular Function in Patients With Refractory Angina and Raised Lipoprotein (a), Treated With Lipoprotein Apheresis
Brief Title: Lipoprotein Apheresis in Refractory Angina Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1880
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Refractory Angina; Raised Lipoprotein(a)>50mg/dL or >500mg/L
Keywords: Refractory Angina; Lipoprotein
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Lipoprotein Apheresis, then sham apheresis (Active Comparator): Three months of weekly lipoprotein apheresis, 1 month washout, then three month sham apheresis
  Interventions: Other: Lipoprotein Apheresis
- First Sham Apheresis, then Lipoprotein Apheresis (Sham Comparator): Three months of weekly sham apheresis, 1 month washout, then three month lipoprotein Apheresis
  Interventions: Other: Sham Apheresis

INTERVENTIONS:
Other: Lipoprotein Apheresis — Weekly lipoprotein apheresis for 3 months
  Arms: First Lipoprotein Apheresis, then sham apheresis
Other: Sham Apheresis — Weekly sham (placebo) apheresis for 3 months
  Arms: First Sham Apheresis, then Lipoprotein Apheresis

SUMMARY:
The goal of this study is to determine the impact of apheresis on clinical parameters and symptoms of patients with refractory angina and raised Lp(a). The investigators will conduct a prospective, randomised controlled crossover study of 20 patients with refractory angina and raised Lp(a), randomised to undergoing lipoprotein apheresis weekly for three months or sham apheresis weekly for three months with assessment of myocardial perfusion, carotid atherosclerosis, endothelial vascular function, thrombogenesis, exercise capacity, angina symptoms and quality of life at the beginning and end of treatment. Patients will then crossover to the opposite study arm with the protocol repeated. The hypothesis is that the above parameters will be improved by lipoprotein apheresis in patients with raised Lp(a) and Refractory Angina. Investigators will also test for the genotypic presence of apolipoprotein(a) gene (LPA) locus variants (rs10455872 and rs3798220) which are thought to be associated with an increased level of Lp(a) and an increased risk of coronary disease.

DETAILED DESCRIPTION:
Angina which is refractory to conventional medical therapy and revascularisation is challenging to manage. Lipoprotein(a) or Lp(a) is a genetically determined form of LDL-cholesterol, elevation of which is an independent risk factor and predictor of adverse cardiovascular events. Lp(a) is felt to increase cardiovascular risk via its prothrombotic effect and by enhancing intimal lipoprotein deposition. Lipoprotein apheresis is the most effective treatment for raised Lp(a). Lipid lowering agents such as statins have little to no effect on Lp(a) levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with refractory angina for more than three months.
* Two or more episodes of angina per week.
* Previous history of myocardial infarction, coronary artery bypass graft (CABG) surgery,percutaneous coronary intervention (PCI) or any combination of the above.
* Prescribed optimal medical therapy.
* Hypercholesterolaemia with an elevated Lp(a) > 50mg/dL and an LDL-cholesterol less than 4.0mmol/L despite optimal lipid lowering drug therapy.

Exclusion Criteria:

* Patients with poor calibre veins for cannulation.
* Patients with any other chronic systemic illness such as liver or renal failure, neoplastic disease, overt cardiac failure, unstable coronary artery disease, coronary revascularisation or a myocardial infarction within the previous eight weeks.
* Pregnancy, untreated diabetes mellitus, untreated arterial hypertension, and those with general contraindications to undergoing Cardiovascular magnetic resonance imaging or contraindications to adenosine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dudley Pennell, MB BChir MA MD FRCP, Principal Investigator — Imperial College London; Mahmoud Barbir, MB BCh, FRCP, Study Director — Royal Brompton and Harfield Hospital, Imperial College
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan TZ, Hsu LY, Arai AE, Rhodes S, Pottle A, Wage R, Banya W, Gatehouse PD, Giri S, Collins P, Pennell DJ, Barbir M. Apheresis as novel treatment for refractory angina with raised lipoprotein(a): a randomized controlled cross-over trial. Eur Heart J. 2017 May 21;38(20):1561-1569. doi: 10.1093/eurheartj/ehx178. PMID 28453721

RESULTS

PARTICIPANT FLOW:
Groups:
- First Lipoprotein Apheresis, Then Sham Apheresis: Three months of weekly lipoprotein apheresis, 1 month of washout then three month of sham apheresis
- First Sham Apheresis, Then Lipoprotein Apheresis: Three months of weekly sham apheresis, 1 month of washout then three months of weekly lipoprotein apheresis
Period: First Intervention
Arm/Group | First Lipoprotein Apheresis, Then Sham Apheresis | First Sham Apheresis, Then Lipoprotein Apheresis
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout
Arm/Group | First Lipoprotein Apheresis, Then Sham Apheresis | First Sham Apheresis, Then Lipoprotein Apheresis
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | First Lipoprotein Apheresis, Then Sham Apheresis | First Sham Apheresis, Then Lipoprotein Apheresis
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participant: Participant were randomised to undergoing lipoprotein apheresis weekly for three months or sham apheresis weekly for three months with assessment of myocardial perfusion, carotid atherosclerosis, endothelial vascular function, thrombogenesis, exercise capacity, angina symptoms and quality of life at the beginning and end of treatment. Patients then crossovered to the opposite study arm with the protocol repeated.
Arm/Group | All Study Participant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Quantitative Myocardial Perfusion Measured by Stress/Rest Cardiovascular Magnetic Resonance Imaging
Description: Baseline compare to 3 month, changes presented Determine the impact of lipoprotein apheresis on quantitative myocardial perfusion measured by stress/rest cardiovascular magnetic resonance imaging.
  Increase means better outcome
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: ratio
Groups:
- Lipoprotein Apheresis: Three months of weekly lipoprotein apheresis
- Sham Apheresis: Three months of weekly sham apheresis
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
ratio | 0.47 [0.31 to 0.63] | -0.16 [-0.33 to 0.02]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Carotid Atherosclerosis/Plaque Burden Determined by Cardiovascular Magnetic Resonance Imaging
Description: Changes from baseline to 3 months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: mm3
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
mm3 | -335 [-423 to -247] | 127 [72 to 183]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Endothelial Vascular Function
Description: EndoPat LnRHI - natural logarithm of reactive hyperaemia index. Increase - better outcome
Time Frame: Within 7 days before and after 3 months of weekly lipoprotein apheresis
Measure: Mean (95% Confidence Interval); unit: index
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
index | -0.05 [-0.08 to 0.19] | -0.03 [-0.18 to 0.11]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.14, t-test, 2 sided

4. Secondary Outcome: Change in Seattle Angina Questionnaire Score
Description: SAQ-Angina stability, increase means improvement. 0-100 scale, Higher score means improvements
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
units on a scale | 17.5 [6.7 to 28.3] | -1.75 [-17.1 to 9.55]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.016, t-test, 2 sided

5. Secondary Outcome: Change in SF-36 Quality of Life Score
Description: Quality of Life score following, 0-100 score, high score improve quality of life
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
units on a scale | 7.5 [5 to 13] | -2 [-4.5 to 1]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Exercise Capacity Determined by Six Minute Walk Test
Description: Six minute walk test, patient can walk longer distance means improvements
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: meter
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
meter | 70.5 [41.5 to 105.5] | 3.5 [-15.1 to 30.8]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Changes in Markers of Thrombogenesis
Description: Thrombogenesis, Reduce value is better to the patients
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
Number analyzed (Participants) | 20 | 20
seconds | -355 [-738 to -88.5] | 36 [-56 to 204]
Statistical Analysis 1: Comparison: Lipoprotein Apheresis vs Sham Apheresis; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lipoprotein Apheresis | Sham Apheresis
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes